CLINICAL TRIAL: NCT06828354
Title: An Open-label, Randomized, Multicenter Phase III Clinical Trial of SHR-A1811 Versus Investigator-selected Chemotherapy for Platinum-resistant Relapsed Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: A Study of SHR-A1811 in Subjects With Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-315
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Gemcitabine; Injections; Topotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 group (Experimental)
  Interventions: Drug: SHR-A1811
- Chemotherapy group (Active Comparator)
  Interventions: Drug: Paclitaxel Injection; Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Topotecan Hydrochloride for Injection

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811.
  Arms: SHR-A1811 group
Drug: Paclitaxel Injection — Paclitaxel Injection.
  Arms: Chemotherapy group
Drug: Doxorubicin Hydrochloride Liposome Injection — Doxorubicin Hydrochloride Liposome Injection.
  Arms: Chemotherapy group
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for Injection.
  Arms: Chemotherapy group
Drug: Topotecan Hydrochloride for Injection — Topotecan Hydrochloride for Injection.
  Arms: Chemotherapy group

SUMMARY:
This is an open-label study to evaluate the safety and efficacy of SHR-A1811 for injection in subjects with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and signed the Informed consent forms (ICF).
2. Measurable disease, as defined by RECIST v1.1.
3. The Eastern Cancer Cooperative Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Symptomatic, untreated or active central nervous system metastases.
2. Have uncontrolled or severe cardiovascular disease.
3. With any active autoimmune disease or history of autoimmune disease.
4. Patients with active hepatitis B or hepatitis C.
5. Severe infections prior to initiation of study treatment.
6. Patients with active tuberculosis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From day 1 to 10 months.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From day 1 to 12 months.
Disease control rate (DCR) | From day 1 to 12 months.
Duration of response (DOR) | From day 1 to 12 months.
Overall survival (OS) | From day 1 to 12 months.
Response rate (RR) | From day 1 to 12 months.
Adverse events (AEs) | From day 1 to 40 days after the last dose.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided